CLINICAL TRIAL: NCT02428140
Title: Post-Embolic Rhythm Detection With Implantable Versus External Monitoring: Pilot and Feasibility Study
Brief Title: Post-Embolic Rhythm Detection With Implantable Versus External Monitoring
Acronym: PERDIEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: University of Calgary (Other); Alberta Innovates Health Solutions (Other); Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 00051629
Record Dates: First submitted 2015-04-23; First posted 2015-04-28 (Estimated); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2021-10

CONDITIONS: Stroke; Atrial Fibrillation; Arrhythmias, Cardiac
Keywords: ischemic stroke; atrial fibrillation; etiologic investigations; secondary prevention; anticoagulation; arrhythmias; embolic stroke, undetermined etiology; implantable loop recorder; external loop recorder
MeSH Terms: conditions — Stroke; Atrial Fibrillation; Arrhythmias, Cardiac; Ischemic Stroke; Embolic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Implanted Loop Recorder (Experimental): long-term implantable ECG (Medtronic Reveal LINQ) coupled with remote monitoring (MyCareLink) for 12 months
  Interventions: Device: Medtronic Reveal LINQ
- External Loop Recorder (Experimental): external event-triggered ECG loop recorder (Sorin Spiderflash-t) for 30 days
  Interventions: Device: Sorin Spiderflash-t

INTERVENTIONS:
Device: Medtronic Reveal LINQ
  Arms: Implanted Loop Recorder
Device: Sorin Spiderflash-t
  Arms: External Loop Recorder

SUMMARY:
The overall aim of this trial is to determine the most cost effective approach to diagnose paroxysmal atrial fibrillation (PAF) following transient ischemic attack (TIA) and stroke.

A summary of the rationale for this study is as follows:

1. Recently completed randomized trials of cardiac monitoring following stroke have established that PAF is more common than previously recognized in cryptogenic stroke.
2. The majority of TIA/stroke patients will have at least one potential stroke mechanism identified by the time etiologic investigations completed.
3. Detecting PAF in patients with strokes with known causes (eg. lacunar and large vessel atherosclerosis) is clinically important since appropriate anticoagulation for AF reduces stroke recurrence in all patients with prior TIA/stroke not just cryptogenic strokes.
4. There are competing technologies for evaluating cardiac rhythm and diagnosing AF but no cost effectiveness data
5. The rates of PAF in strokes with known causes (SKC) have not been well characterized.

PER-DIEM is a pilot study to compare two different cardiac monitoring technologies as first-line investigations to detect PAF in patients with recent stroke and TIA. The study will also assess whether a pivotal trial is feasible and warranted.

The principal research questions to be addressed in this study will be:

1. Whether implantable loop recorder (ILR) plus remote monitoring will diagnose more paroxysmal AF / atrial flutter and provide a better assessment of the total burden of AF resulting in a greater proportion of patients started on an OAC versus the external loop recorder (ELR) strategy.
2. What is the relative cost-effectiveness as a first-line investigation of long-term implantable ECG (ILR) coupled with remote monitoring for 12 months compared to external event-triggered ECG loop recorder (ELR) for 30 days in the diagnosis clinically actionable AF in following TIA/stroke.

2) What is the feasibility, patient compliance, diagnostic accuracy and rates of AF detection (>30 seconds) of ILR compared to the ELR strategies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of the index event* made by a stroke specialist of an acute ischemic stroke or TIA occurring within the previous 90 days. The event must be either:

  1. an arterial ischemic stroke confirmed by neuroimaging; or
  2. transient ischemic attack with diffusion weighted positive lesion on MRI
* At least one 12-lead ECG has already been obtained as part of the routine clinical post-stroke/TIA work-up, and no ECGs have shown any episodes of atrial fibrillation or atrial flutter
* The patient is being actively investigated for the etiology of the stroke/TIA event and additional cardiac monitoring is desired to screen further for the possibility of occult paroxysmal atrial fibrillation/flutter
* Age 18 years or older
* Informed consent from the patient
* The patient is expected to survive at least 6 months.

Exclusion Criteria:

* Any previously documented atrial fibrillation or atrial flutter, i.e. a past history of atrial fibrillation/flutter or atrial fibrillation/flutter detected on ECG, Holter, or telemetry following the index stroke/TIA event (a remote history of transient perioperative atrial fibrillation is not exclusionary)
* Planned carotid endarterectomy or carotid artery stenting within 90 days
* Any condition for which there is already an indication for long term anticoagulation Pacemaker or implantable cardioverter defibrillator device
* Work-up for stroke that has already included extended (>48 hour) external ECG (excluding telemetry)
* Stroke and/or comorbid illness will prevent completion of planned follow-up assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian H Buck, MD, MSc, Principal Investigator — University of Alberta
Locations (3):
- Canada (3):
  - Foothills Medical Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Grey Nuns Community Hospital, Edmonton, Alberta

REFERENCES:
- [Result] Buck BH, Hill MD, Quinn FR, Butcher KS, Menon BK, Gulamhusein S, Siddiqui M, Coutts SB, Jeerakathil T, Smith EE, Khan K, Barber PA, Jickling G, Reyes L, Save S, Fairall P, Piquette L, Kamal N, Chew DS, Demchuk AM, Shuaib A, Exner DV. Effect of Implantable vs Prolonged External Electrocardiographic Monitoring on Atrial Fibrillation Detection in Patients With Ischemic Stroke: The PER DIEM Randomized Clinical Trial. JAMA. 2021 Jun 1;325(21):2160-2168. doi: 10.1001/jama.2021.6128. PMID 34061146

RESULTS

PARTICIPANT FLOW:
Groups:
- Implanted Loop Recorder: long-term implantable ECG (Medtronic Reveal LINQ) coupled with remote monitoring (MyCareLink) for 12 months
  Medtronic Reveal LINQ
- External Loop Recorder: external event-triggered ECG loop recorder (Sorin Spiderflash-t) for 30 days
  Sorin Spiderflash-t
Period: Overall Study
Arm/Group | Implanted Loop Recorder | External Loop Recorder
Started | 150 | 150
Completed | 150 | 150
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Implanted Loop Recorder | External Loop Recorder | Total
Number analyzed (Participants) | 150 | 150 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 150 | 150 | 300
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65.5 [58.1 to 73.7] | 63.4 [54.7 to 73.5] | 64.2 [56.1 to 73.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 60 | 121
  Male | 89 | 90 | 179
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race/ethnicity data was not collected.
Region of Enrollment [Number; unit: participants]
  Canada | 150 | 150 | 300
Hypertension [Count of Participants; unit: Participants] | 93 | 94 | 187
Previous Stroke [Count of Participants; unit: Participants] | 36 | 34 | 70

OUTCOME MEASURES:

1. Primary Outcome: Definite AF or Highly Probable AF
Description: Definite AF or highly probable AF (adjudicated new AF lasting ≥2 minutes within 12 months of randomization)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Implanted Loop Recorder | External Loop Recorder
Number analyzed (Participants) | 150 | 150
Participants | 23 | 7
Statistical Analysis 1: Comparison: Implanted Loop Recorder vs External Loop Recorder; Test type: Superiority; p = 0.003, t-test, 2 sided; Risk Ratio (RR) = 3.29, 95% CI 2-sided [1.45 to 7.42]

2. Secondary Outcome: AF Lasting ≥2 Min or Death by 12 Months
Description: Detection of atrial fibrillation lasting ≥ 2 minutes or death by 12 months.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Implanted Loop Recorder | External Loop Recorder
Number analyzed (Participants) | 150 | 150
Participants | 26 | 10
Statistical Analysis 1: Comparison: Implanted Loop Recorder vs External Loop Recorder; Test type: Superiority; p = .005, t-test, 2 sided; Risk Difference (RD) = 10.7, 95% CI 2-sided [3.4 to 17.9]

3. Secondary Outcome: TIA
Description: Transient ischemic attack.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Implanted Loop Recorder | External Loop Recorder
Number analyzed (Participants) | 150 | 150
Participants | 6 | 2
Statistical Analysis 1: Comparison: Implanted Loop Recorder vs External Loop Recorder; Test type: Superiority; p = 0.28, t-test, 2 sided; Risk Difference (RD) = 2.7, 95% CI 2-sided [-1.0 to 6.3]

4. Secondary Outcome: Recurrent Stroke
Description: Recurrent ischemic stroke.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Implanted Loop Recorder | External Loop Recorder
Number analyzed (Participants) | 150 | 150
Participants | 5 | 8

5. Secondary Outcome: Hemorrhage
Description: Intracerebral hemorrhage.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Implanted Loop Recorder | External Loop Recorder
Number analyzed (Participants) | 150 | 150
Participants | 1 | 1
Statistical Analysis 1: Comparison: Implanted Loop Recorder vs External Loop Recorder; Test type: Superiority; Risk Difference (RD) = 0, 95% CI 2-sided [-1.8 to 1.8]

6. Secondary Outcome: Death
Description: Participant death.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Implanted Loop Recorder | External Loop Recorder
Number analyzed (Participants) | 150 | 150
Participants | 3 | 3
Statistical Analysis 1: Comparison: Implanted Loop Recorder vs External Loop Recorder; Test type: Superiority; Risk Difference (RD) = 0, 95% CI 2-sided [-3.2 to 3.2]

7. Secondary Outcome: Oral Anticoagulation Therapy
Description: Initiation of oral anticoagulation therapy in patients with definite AF.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Implanted Loop Recorder | External Loop Recorder
Number analyzed (Participants) | 150 | 150
Participants | 23 | 7

8. Secondary Outcome: ≥1 Serious Adverse Event
Description: Patients with ≥1 serious adverse event.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Implanted Loop Recorder | External Loop Recorder
Number analyzed (Participants) | 150 | 150
Participants | 14 | 4

9. Secondary Outcome: Compliance
Description: Compliance with assigned therapy (accept ILR, conduct at least 80% of ELR assessments)
Time Frame: 12 months
Population: Outcome measure not performed.
Arm/Group | Implanted Loop Recorder | External Loop Recorder
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Costs of Cardiac and Non-cardiac Investigations
Description: Costs for all cardiac and non-cardiac investigations related to etiologic workup of index stroke / TIA.
Time Frame: 12 months
Population: Outcome measure not performed.
Arm/Group | Implanted Loop Recorder | External Loop Recorder
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Duration of Any Detected Atrial Fibrillation / Atrial Flutter.
Description: Total duration of any detected atrial fibrillation / atrial flutter.
Time Frame: 12 months
Population: Outcome measure not performed.
Arm/Group | Implanted Loop Recorder | External Loop Recorder
Number analyzed (Participants) | 0 | 0

12. Other Pre Specified Outcome: Predictors of AF Detection
Description: Association between baseline clinical characteristics (e.g. comorbidities, burden of supraventricular ectopy on Holter, left atrial dimension) and subsequent detection of AF
Time Frame: 12 months
Population: Outcome measure not performed
Arm/Group | Implanted Loop Recorder | External Loop Recorder
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Description: A clinical events committee reviewed all serious adverse events 12 months after study initiation to ensure that neither group had a disproportionate accumulation of adverse events. The study used approved devices therefore nonserious adverse events were not tracked.
Arm/Group | Implanted Loop Recorder | External Loop Recorder
All-Cause Mortality (participants affected / at risk) | 3/150 | 3/150
Serious Adverse Events (participants affected / at risk) | 14/150 | 4/150
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Implanted Loop Recorder (N=150) | External Loop Recorder (N=150)
Bacterial peritonitis (Infections and infestations) | 1 | 0
Bladder Neck Obstruction (Renal and urinary disorders) | 1 | 0
Cardiac Amyloidosis (Cardiac disorders) | 1 | 0
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Device-Related Skin Erosion (Skin and subcutaneous tissue disorders) | 1 | 0
Femoral fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 | 0
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
High-Grade Symptomatic Atrioventricular Block (Cardiac disorders) | 1 | 0
Hip Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 2
Pancolitis (Gastrointestinal disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Multiple Trauma (Musculoskeletal and connective tissue disorders) | 1 | 0
Quadriceps Tendon Rupture (Musculoskeletal and connective tissue disorders) | 1 | 0
Recrudescence of Stroke Deficits (Nervous system disorders) | 1 | 0
Renal Colic (Renal and urinary disorders) | 1 | 0
Symptomatic Sinus Bradycardia (Cardiac disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-02-22): https://cdn.clinicaltrials.gov/large-docs/40/NCT02428140/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT02428140/SAP_001.pdf